CLINICAL TRIAL: NCT00296686
Title: A Pilot Study of Treatment for Refractory Depression With Sequential Trials of Tranylcypromine, Tranylcypromine Plus Dextroamphetamine, Tranylcypromine Plus Triiodothyronine.
Brief Title: Sequential Tranylcypromine (TC), TC + Dextroamphetamine and TC + Triiodothyronine for Refractory Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study is no longer funded.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #4213; NCT00296686 (Other Grant/Funding Number: There is no grantor or funder)
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Major Depression
Keywords: Major Depression; Refractory Depression; Tranylcypromine; Dextroamphetamine; Triiodothyronine
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Tranylcypromine; Dextroamphetamine; Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tranylcypromine (Experimental): sequential tranylcypromine (TC) followed by TC + dextroamphetamine followed by TC + T3
  Interventions: Drug: Tranylcypromine; Drug: Dextroamphetamine; Drug: Triiodothyronine

INTERVENTIONS:
Drug: Tranylcypromine — standard dose:60 mg/d for a minimum of 8 weeks, a maximum of 17 weeks; high dose for non-remitters: up to 120 mg/day for a maximum of 9 weeks.
  Other Names: Parnate
Drug: Dextroamphetamine — up to 40 mg/day for 9 weeks, in combination with high dose of tranylcypromine for patients not remitting on the standard or high doses of tranylcypromine alone.
  Other Names: Dexedrine
Drug: Triiodothyronine — For patients not remitting on higher dose of tranylcypromine plus dextroamphetamine: Up to 75 mg/day for 8 weeks(+/- dextroamphetamine) (max 8 weeks) in combination with highest does of tranylcypromine (up to 120mg/day).
  Other Names: Cytomel

SUMMARY:
This pilot study will assess the efficacy of several sequential pharmacological treatments for patients with Refractory Depression.

DETAILED DESCRIPTION:
This pilot study will recruit 40 patients with Major Depression and a history of at least two failed prior adequate somatic treatments. In addition to usual physical work-up, all patients will have extensive thyroid testing, and then will receive standard dose Tranylcypromine (i.e., max. 60 mg/d). Non-remitters will have dose increased to max. 120 mg/d if tolerated. Non-remitters to high dose Tranylcypromine will then have Dextroamphetamine added with frequent blood pressure monitoring to max. 40 mg/d. Non-remitters will have Triiodothyronine added to the Tranylcypromine.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-65
* Major Depression
* At least two prior ineffective antidepressant trials (at least 2 different mechanisms) or 1 inadequate ECT trial (at least 8 bilateral treatments)
* Physically healthy

Exclusion Criteria:

* Known Tranylcypromine allergy
* Unable to follow tyramine-free diet
* Known allergy, intolerance or prior addiction to any stimulant would preclude patient's inclusion in the Dextroamphetamine portion of the protocol
* Current substance use disorder including alcohol)(past six months); ever dependent on stimulants would preclude Dextroamphetamine portion of the protocol
* Unable or unwilling to discontinue antidepressants including OTC antidepressants such as St. John's Wort
* History of psychosis, such as schizophrenia or psychotic depression; history of bipolar mania will be allowed if on adequate mood stabilizer
* Suicidal ideation/activity that makes outpatient treatment unsafe, unless protocol can be conducted as inpatient
* Current systolic BP > 149 or diastolic BP > 89 mm Hg (two readings); adequately treated hypertension is acceptable
* Evidence of hypo- or hyperthyroidism
* Pregnancy, lactation, refusal to use adequate birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | up to 10 mos.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | up to 10 mos.
Clinical Global Impression (CGI) | up to 10 mos.
Patient Global Impression (PGI) | up to 10 mos.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Stewart, MD, Principal Investigator — New York State Psychiatric Institute - Columbia University Department of Psychiatry
Locations (1):
- Depression Evaluation Service - New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Stewart JW, Deliyannides DA, McGrath PJ. How treatable is refractory depression? J Affect Disord. 2014;167:148-52. doi: 10.1016/j.jad.2014.05.047. Epub 2014 Jun 4. PMID 24972362
- See also: Depression Evaluation Service - official website — http://www.depression-nyc.org
- See also: New York State Psychiatric Institute - official website — http://www.nyspi.org